CLINICAL TRIAL: NCT01779362
Title: Restoring Insulin Secretion Adult Medication Study
Brief Title: RISE Adult Medication Study
Acronym: RISE Adult
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RISE Study Group (Network)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RISE Adult; 5U01DK094406-02 (NIH)
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2018-08

CONDITIONS: Prediabetes; Type 2 Diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Metformin; Liraglutide; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Metformin alone (Active Comparator): Metformin will be titrated to the maximum dose tolerated (up to 2000 mg/day). Participants randomized to the metformin-alone arm will be blinded to treatment.
  Interventions: Drug: Metformin
- Glargine followed by Metformin (Active Comparator): Basal insulin glargine for 3 months titrated to achieve a morning fasting blood glucose of 80-90 mg/dl, followed by open-label metformin (titrated up to 2000 mg/day) for 9 months.
  Interventions: Drug: Metformin; Drug: Glargine
- Placebo (Placebo Comparator): Placebo - masked to metformin-alone. Placebo will be titrated to the maximum number of tablets equivalent to maximum dose of metformin.
  Interventions: Drug: Placebo
- Liraglutide + Metformin (Active Comparator): Liraglutide + open-label Metformin. Liraglutide will be titrated to the maximum dose tolerated (up to 1.8 mg/day) after which metformin will be titrated to the maximum dose tolerated (up to 2000 mg/day).
  Interventions: Drug: Metformin; Drug: Liraglutide

INTERVENTIONS:
Drug: Metformin — Titrated to 1000 mg BID
  Other Names: Glucophage
  Arms: Glargine followed by Metformin; Liraglutide + Metformin; Metformin alone
Drug: Liraglutide — Titrated to 1.8 mg/day
  Other Names: Victoza
  Arms: Liraglutide + Metformin
Drug: Glargine — Titrated to target fasting glucose <90 mg/dl
  Other Names: Insulin glargine, Lantus
  Arms: Glargine followed by Metformin
Drug: Placebo — Matching to metformin 1000 mg BI
  Arms: Placebo

SUMMARY:
The RISE Adult Medication Study is a 4-arm, 3-center, clinical trial of adults with prediabetes and early type 2 diabetes to address the hypothesis that aggressive glucose lowering will lead to recovery of beta-cell function that will be sustained after withdrawal of treatment. Adult participants (ages 20-65) will be randomized to one of the following treatment regimens: (1) blinded placebo, (2) blinded metformin alone, (3) early intensive insulin treatment with basal insulin glargine followed by open-label metformin, (4) the glucagon-like peptide-1 receptor agonist (GLP-1RA) liraglutide plus open-label metformin.

The primary clinical question RISE will address is: Are improvements in ß-cell function following 12 months of active treatment maintained for 3 months following the withdrawal of therapy? Secondary outcomes will assess durability of glucose tolerance following withdrawal of therapy, and whether biomarkers obtained in the fasting state predict parameters of ß-cell function, insulin sensitivity and glucose tolerance and the response to an intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting plasma glucose 95-125 mg/dl plus 2-hour glucose ≥140 mg/dl on 75 gm OGTT plus HbA1c ≤7.0%. There is no upper limit for the 2-hour glucose on OGTT.
2. Age 20-65 years
3. Body mass index (BMI) ≥25 kg/m2 but ≤50 kg/m2
4. Self-reported diabetes <1 year in duration
5. Drug naïve (no prior to oral glucose lowering agent(s), insulin or other injectable glucose lowering agents)

Exclusion Criteria:

1. Underlying disease likely to limit life span and/or increase risk of intervention or an underlying condition that is likely to limit ability to participate in outcomes assessment
2. An underlying disease that affects glucose metabolism other than type 2 diabetes
3. Taking medications that affect glucose metabolism, or has an underlying condition that is likely to require such medications
4. Active infections
5. Renal disease (serum creatinine >1.4 mg/dl for men; >1.3 mg/dl for women) or serum potassium abnormality (<3.4 or >5.5 mmol/l)
6. Anemia (hemoglobin <11 g/dl in women, <12 g/dl in men) or known coagulopathy
7. Cardiovascular disease, including uncontrolled hypertension. Participants must be able to safely tolerate administration of intravenous fluids required during clamp studies.
8. History of conditions that may be precipitated or exacerbated by a study drug:

   1. Pancreatitis
   2. Serum alanine transaminase (ALT) more than 3 times the upper limit of normal
   3. Excessive alcohol intake
   4. Suboptimally treated thyroid disease
   5. Medullary carcinoma of the thyroid or MEN-2 (in participant or a family history)
   6. Hypertriglyceridemia (>400 mg/dl despite treatment)
9. Conditions or behaviors likely to affect the conduct of the RISE Study

   1. Unable or unwilling to give informed consent
   2. Unable to adequately communicate with clinic staff
   3. Another household member is a participant or staff member in RISE
   4. Current, recent or anticipated participation in another intervention research project that would interfere with any of the interventions/outcomes in RISE
   5. Weight loss of >5% in past three months for any reason other than post-partum weight loss. Participants taking weight loss drugs or using preparations taken for intended weight loss are excluded.
   6. Likely to move away from participating clinics in next two years
   7. Women of childbearing potential who are unwilling to use adequate contraception
   8. Current (or anticipated) pregnancy and lactation.
   9. Major psychiatric disorder that, in the opinion of clinic staff, would impede the conduct of RISE
10. Additional conditions may serve as criteria for exclusion at the discretion of the local site.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2013-04; Primary Completion 2019-02 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available through the NIDDK repository within 2 years after the final participant visit. Data can be obtained from the NIDDK repository.

REFERENCES:
- [Background] RISE Consortium. Restoring Insulin Secretion (RISE): design of studies of beta-cell preservation in prediabetes and early type 2 diabetes across the life span. Diabetes Care. 2014;37(3):780-8. doi: 10.2337/dc13-1879. Epub 2013 Nov 5. PMID 24194506
- [Background] Hannon TS, Kahn SE, Utzschneider KM, Buchanan TA, Nadeau KJ, Zeitler PS, Ehrmann DA, Arslanian SA, Caprio S, Edelstein SL, Savage PJ, Mather KJ; RISE Consortium. Review of methods for measuring beta-cell function: Design considerations from the Restoring Insulin Secretion (RISE) Consortium. Diabetes Obes Metab. 2018 Jan;20(1):14-24. doi: 10.1111/dom.13005. Epub 2017 Jun 22. PMID 28493515
- [Derived] Tjaden AH, Edelstein SL, Arslanian S, Barengolts E, Caprio S, Cree-Green M, Lteif A, Mather KJ, Savoye M, Xiang AH, Kahn SE. Reproducibility of Glycemic Measures Among Dysglycemic Youth and Adults in the RISE Study. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1125-e1133. doi: 10.1210/clinem/dgad135. PMID 36938582
- [Derived] Utzschneider KM, Ehrmann DA, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Edelstein SL, Hannon TS, Kahn SE, Kozedub A, Mather KJ, Nadeau KJ, Sam S, Tripputi M, Xiang AH, El Ghormli L; RISE Consortium. Weight loss and beta-cell responses following gastric banding or pharmacotherapy in adults with impaired glucose tolerance or type 2 diabetes: a randomized trial. Obesity (Silver Spring). 2022 Aug;30(8):1579-1588. doi: 10.1002/oby.23475. PMID 35894078
- [Derived] Utzschneider KM, Tripputi MT, Kozedub A, Barengolts E, Caprio S, Cree-Green M, Edelstein SL, El Ghormli L, Hannon TS, Mather KJ, Palmer J, Nadeau KJ; RISE Consortium. Differential loss of beta-cell function in youth vs. adults following treatment withdrawal in the Restoring Insulin Secretion (RISE) study. Diabetes Res Clin Pract. 2021 Aug;178:108948. doi: 10.1016/j.diabres.2021.108948. Epub 2021 Jul 15. PMID 34274407
- [Derived] Kahn SE, Edelstein SL, Arslanian SA, Barengolts E, Caprio S, Ehrmann DA, Hannon TS, Marcovina S, Mather KJ, Nadeau KJ, Utzschneider KM, Xiang AH, Buchanan TA; RISE Consortium; Rise Consortium Investigators:. Effect of Medical and Surgical Interventions on alpha-Cell Function in Dysglycemic Youth and Adults in the RISE Study. Diabetes Care. 2021 Sep;44(9):1948-1960. doi: 10.2337/dc21-0461. Epub 2021 Jun 16. PMID 34135015
- [Derived] Sam S, Edelstein SL, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Ehrmann DA, Hannon TS, Tjaden AH, Kahn SE, Mather KJ, Tripputi M, Utzschneider KM, Xiang AH, Nadeau KJ; RISE Consortium; RISE Consortium Investigators. Baseline Predictors of Glycemic Worsening in Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes in the Restoring Insulin Secretion (RISE) Study. Diabetes Care. 2021 Sep;44(9):1938-1947. doi: 10.2337/dc21-0027. Epub 2021 Jun 15. PMID 34131048
- [Derived] Kahn SE, Mather KJ, Arslanian SA, Barengolts E, Buchanan TA, Caprio S, Ehrmann DA, Hannon TS, Marcovina S, Nadeau KJ, Utzschneider KM, Xiang AH, Edelstein SL; RISE Consortium; Rise Consortium Investigators:. Hyperglucagonemia Does Not Explain the beta-Cell Hyperresponsiveness and Insulin Resistance in Dysglycemic Youth Compared With Adults: Lessons From the RISE Study. Diabetes Care. 2021 Sep;44(9):1961-1969. doi: 10.2337/dc21-0460. Epub 2021 Jun 15. PMID 34131047
- [Derived] Arslanian SA, El Ghormli L, Kim JY, Tjaden AH, Barengolts E, Caprio S, Hannon TS, Mather KJ, Nadeau KJ, Utzschneider KM, Kahn SE; RISE Consortium. OGTT Glucose Response Curves, Insulin Sensitivity, and beta-Cell Function in RISE: Comparison Between Youth and Adults at Randomization and in Response to Interventions to Preserve beta-Cell Function. Diabetes Care. 2021 Mar;44(3):817-825. doi: 10.2337/dc20-2134. Epub 2021 Jan 12. PMID 33436401
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] RISE Consortium. Obesity and insulin sensitivity effects on cardiovascular risk factors: Comparisons of obese dysglycemic youth and adults. Pediatr Diabetes. 2019 Nov;20(7):849-860. doi: 10.1111/pedi.12883. Epub 2019 Jul 29. PMID 31301210
- [Derived] RISE Consortium. Lack of Durable Improvements in beta-Cell Function Following Withdrawal of Pharmacological Interventions in Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes. Diabetes Care. 2019 Sep;42(9):1742-1751. doi: 10.2337/dc19-0556. Epub 2019 Jun 9. PMID 31178434
- [Derived] RISE Consortium; RISE Consortium Investigators. Effects of Treatment of Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes With Metformin Alone or in Combination With Insulin Glargine on beta-Cell Function: Comparison of Responses In Youth And Adults. Diabetes. 2019 Aug;68(8):1670-1680. doi: 10.2337/db19-0299. Epub 2019 Jun 9. PMID 31178433
- [Derived] RISE Consortium. Metabolic Contrasts Between Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes: II. Observations Using the Oral Glucose Tolerance Test. Diabetes Care. 2018 Aug;41(8):1707-1716. doi: 10.2337/dc18-0243. Epub 2018 Jun 25. PMID 29941498
- [Derived] RISE Consortium. Metabolic Contrasts Between Youth and Adults With Impaired Glucose Tolerance or Recently Diagnosed Type 2 Diabetes: I. Observations Using the Hyperglycemic Clamp. Diabetes Care. 2018 Aug;41(8):1696-1706. doi: 10.2337/dc18-0244. Epub 2018 Jun 25. PMID 29941497

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin
Started | 65 | 67 | 67 | 68
Completed | 56 | 65 | 58 | 53
Not Completed | 9 | 2 | 9 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin | Total
Number analyzed (Participants) | 65 | 67 | 67 | 68 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (8.2) | 53.5 (9.3) | 52.8 (10.0) | 54.0 (8.1) | 53.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 23 | 25 | 29 | 114
  Male | 28 | 44 | 42 | 39 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 34 | 37 | 30 | 40 | 141
  Race/Ethnicity: Black | 19 | 21 | 21 | 20 | 81
  Race/Ethnicity: Hispanic | 6 | 5 | 11 | 6 | 28
  Race/Ethnicity: All other | 6 | 4 | 5 | 2 | 17
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.0 (5.1) | 35.0 (5.9) | 34.4 (5.9) | 35.6 (5.8) | 35.0 (5.7)
HbA1c [Mean (Standard Deviation); unit: % of glycosylated hemoglobin] | 5.77 (0.40) | 5.80 (0.33) | 5.73 (0.43) | 5.69 (0.39) | 5.75 (0.39)
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] | 6.21 (0.67) | 6.22 (0.74) | 6.08 (0.58) | 6.11 (0.50) | 6.15 (0.63)
2-hour OGTT glucose [Mean (Standard Deviation); unit: mmol/L] | 10.1 (2.4) | 10.3 (2.4) | 10.1 (2.3) | 9.9 (2.2) | 10.1 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: ß-cell Response Measured by Hyperglycemic Clamp
Description: Clamp measures of ß-cell response, co-primary outcomes
Time Frame: 3-months after medication washout (Month 15)
Population: Primary analysis was on all participants who attended their M15 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin
Number analyzed (Participants) | 56 | 65 | 58 | 53
nmol/L
  Steady State C-peptide | 3.65 [1.94 to 6.87] | 3.58 [1.68 to 8.33] | 3.60 [1.72 to 7.53] | 3.73 [1.87 to 7.44]
  ACPRmax | 4.61 [2.00 to 10.66] | 4.32 [1.58 to 11.80] | 4.45 [1.56 to 12.71] | 4.58 [2.21 to 9.48]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin vs Placebo vs Liraglutide + Metformin; Seemingly unrelated regression was used to compare treatment arms on the combination of insulin sensitivity (M/I as calculated from the hyperglycemic clamp) and insulin secretion (steady-state C-peptide and ACPRmax as co-primary; ACPRg as major secondary,). See statistical analysis plan for further details and R code; Test type: Superiority; p > 0.05, Regression, Linear — All analyses were conducted with values on a log scale and re-exponentiated for presentation; Measures of ß-cell response were modeled simultaneously with insulin sensitivity (M/I) using 2-df seemingly unrelated regression models

2. Primary Outcome: Insulin Sensitivity, M/I
Description: Clamp measure of insulin sensitivity
Time Frame: 3-months after a medication washout
Population: All participants with a Month 15 visit
Measure: Geometric Mean (95% Confidence Interval); unit: x 10-5 mmol/kg/min per pmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin
Number analyzed (Participants) | 56 | 65 | 58 | 53
x 10-5 mmol/kg/min per pmol/L | 3.53 [0.67 to 18.49] | 3.38 [0.61 to 18.84] | 3.63 [0.95 to 13.84] | 3.49 [0.90 to 13.54]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin vs Placebo vs Liraglutide + Metformin; Test type: Superiority; p > 0.05, Regression, Linear

3. Secondary Outcome: ACPRg
Description: First phase response from the hyperglycemic clamp
Time Frame: 3-months after a medication washout
Population: Analysis was on all participants able to have a M15 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin
Number analyzed (Participants) | 56 | 65 | 58 | 53
nmol/L | 1.68 [0.84 to 3.34] | 1.68 [0.91 to 3.09] | 1.68 [0.86 to 3.26] | 1.68 [0.99 to 2.83]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin vs Placebo vs Liraglutide + Metformin; Test type: Superiority; p > 0.05, Regression, Linear

4. Secondary Outcome: ß-cell Function Measured by Hyperglycemic Clamp Techniques at M12
Description: Participants had 12-months of active therapy. Secondary results at the end of active intervention.
Time Frame: Secondary analysis was on all participants with a Month 12 visit.
Population: Secondary analysis was on all participants with a Month 12 visit.
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin
Number analyzed (Participants) | 56 | 65 | 58 | 53
nmol/L
  ACRPg | 1.93 [1.09 to 3.40] | 1.88 [1.06 to 3.22] | 1.69 [0.89 to 3.22] | 2.68 [1.28 to 5.60]
  Steady State C-peptide | 11.7 [5.6 to 24.3] | 11.6 [5.6 to 24.3] | 10.8 [5.1 to 22.7] | 21.2 [9.3 to 48.3]
  ACRPmax | 13.4 [5.9 to 30.7] | 14.1 [5.8 to 34.3] | 13.6 [5.1 to 36.1] | 10.1 [3.5 to 28.5]
Statistical Analysis 1: Comparison: Metformin Alone vs Glargine Followed by Metformin vs Placebo vs Liraglutide + Metformin; Analyses were completed on a log scale and re-exponentiated for display; Test type: Superiority; p < 0.001, ANOVA — For all 3 secondary outcomes at M12, p<0.001, with the Liraglutide+Metformin group different from the 3 others (all p<0.001)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Metformin Alone | Glargine Followed by Metformin | Placebo | Liraglutide + Metformin
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/67 | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 5/65 | 2/67 | 3/67 | 7/68
Other Adverse Events (participants affected / at risk) | 29/65 | 28/67 | 23/67 | 30/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Alone (N=65) | Glargine Followed by Metformin (N=67) | Placebo (N=67) | Liraglutide + Metformin (N=68)
Chest pain (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) — Hospital admission for chest pain
Kidney Stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Kidney Stone Removal
Spinal decompression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Elective spinal decompression surgery
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Motor vehicle accident w/head injury
Cholelithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Cholelithiasis/ Cholecystitis
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hospitalization for pain control related to chronic back pain
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Sepsis due to scalp cellulitis
Arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left knee total arthroplasty
Food poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for food poisoning
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for pneumonia, bronchitis, respiratory infection
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for earaches and numbness
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Surgical relief of carpal tunnel nerve pain
Reduced ability to walk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hospitalization due to diminishing ability to support weight and ambulate
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hospitalization for asthma attack
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Foot surgery for arthritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Alone (N=65) | Glargine Followed by Metformin (N=67) | Placebo (N=67) | Liraglutide + Metformin (N=68)
Any low blood sugar (Endocrine disorders) | 3 (3) | 8 (8) | 5 (5) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6) | 4 (4) | 1 (1)
GI Symptoms (Gastrointestinal disorders) | 23 (23) | 12 (12) | 10 (10) | 28 (28)
Diabetes symptoms (Endocrine disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT01779362/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT01779362/SAP_001.pdf